CLINICAL TRIAL: NCT06178848
Title: Comparison of Quantitative EEG Parameters During Anesthesia Emergence Between Remimazolam Group and Propofol Group
Brief Title: EEG Parameters Between Remimazolam- and Propofol-based Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2022-1405
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Cholecystitis, Acute; Gallbladder Neoplasms; Acalculous Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute; Gallbladder Neoplasms; Acalculous Cholecystitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The principal investigator and the anesthesiologist directly involved in anesthetizing the respective patients should be aware of patient allocation due to the nature of research design and anesthesia maintenance. Two research personnel, who are unaware of the type of test drug (blinding), are not involved in anesthesia but are responsible only for data collection and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): During induction, the propofol group initiates with a target-controlled infusion (TCI) of propofol, starting at an effect site concentration of 4.0 ng/ml. After intubation, it is adjusted to maintain an appropriate depth of anesthesia based on the EEG (psi target 40).
  Interventions: Drug: propofol group
- remimazolam group (Experimental): The remimazolam group begins with a continuous infusion of remimazolam at 6 mg/kg/hr, which is then adjusted to 1 mg/kg/hr after loss of consciousness to maintain an appropriate depth of anesthesia based on the EEG (psi target 40).
  Interventions: Drug: remimazolam group

INTERVENTIONS:
Drug: propofol group — During induction, the propofol group initiates with a target-controlled infusion (TCI) of propofol, starting at an effect site concentration of 4.0 ng/ml. After intubation, it is adjusted to maintain an appropriate depth of anesthesia based on the EEG (psi target 40).
  Arms: propofol group
Drug: remimazolam group — The remimazolam group begins with a continuous infusion of remimazolam at 6 mg/kg/hr, which is then adjusted to 1 mg/kg/hr after loss of consciousness to maintain an appropriate depth of anesthesia based on the EEG (psi target 40).
  Arms: remimazolam group

SUMMARY:
This is an observational study comparing perioperative quantitative EEG parameters between the conventional propofol/remifentanil and remimazolam/remifentanil. We aim to compare and analyze the differences in EEG patterns during the postoperative recovery in a group that underwent remimazolam and remifentanil-based total intravenous anesthesia(TIVA), in comparison to propofol and remifentanil-based TIVA

ELIGIBILITY:
Inclusion Criteria:

Patients aged 19 to 65 years who meet the American Society of Anesthesiologists (ASA) physical status classification 1-3 and undergo laparoscopic cholecystectomy at Severance Hospital.

Exclusion Criteria:

Pregnant women, individuals with arrhythmias, emergency surgeries, obesity (BMI > 30), day-surgery, foreigners, and illiterate individuals.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
frontal spectral power | immediately after awakening at the end of the anesthesia, at post-anesthesia care unit (PACU)
  Frontal spectral power in EEG (Electroencephalography) refers to the measurement of electrical activity in the frontal lobes of the brain across different frequency bands. Frontal spectral power specifically focuses on the electrical activity in the frontal region of the brain within these frequency bands. Different frequency bands are associated with different states of brain activity. For example, alpha waves are often associated with relaxation or idling of the brain, while beta waves are linked to more active cognitive processing.

SECONDARY OUTCOMES:
Riker sedation-agitation score | immediately after awakening at the end of the anesthesia, at post-anesthesia care unit (PACU)
  The Richmond Agitation-Sedation Scale (RASS) is a medical assessment tool used to measure a patient's level of agitation or sedation. The Richmond Agitation-Sedation Scale typically ranges from -5 to +4, with each level representing a specific state of sedation or agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, Principal Investigator — Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee Y, Park S, Kim H, Park Y, Lee U, Kwon J, Koo BN, Moon JY. Electroencephalogram Correlates of Delayed Emergence After Remimazolam-Induced Anesthesia Compared to Propofol. Anesth Analg. 2025 Apr 25. doi: 10.1213/ANE.0000000000007516. Online ahead of print. PMID 40279265